CLINICAL TRIAL: NCT05936307
Title: Modulation of Auditory Externalization Abilities by Transcranial Stimulation of the Brain Area Specifically Involved
Brief Title: Externalization and Stimulation
Acronym: STUPEFIX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-A00452-43
Record Dates: First submitted 2023-06-16; First posted 2023-07-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-06

CONDITIONS: Healthy Participants
Keywords: externalization; auditory processing; reality-monitoring; stimulation; HD-TDCS

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized crossover study including 30 healthy participants who will receive active and placebo HD-tDCS in a counterbalanced order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and experimenters (including tDCS operator) will not be informed about the nature (active or placebo) of the stimulation they will receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15 healthy participants active then placebo (Active Comparator): 15 healthy participants will receive a session of active HD-tDCS and then a session of placebo HD-tDCS.
  Interventions: Procedure: High-definition transcranial direct current (HD-tDCS), active condition; Procedure: High-definition transcranial direct current (HD-tDCS), placebo condition
- 15 healthy participants placebo then active (Placebo Comparator): 15 healthy participants will receive a session of placebo HD-tDCS and then a session of active HD-tDCS.
  Interventions: Procedure: High-definition transcranial direct current (HD-tDCS), active condition; Procedure: High-definition transcranial direct current (HD-tDCS), placebo condition

INTERVENTIONS:
Procedure: High-definition transcranial direct current (HD-tDCS), active condition — Participants will receive a session of active HD-tDCS at a current intensity of 2 mA for a duration of 25min. The placement of electrodes will be determined to specifically target the brain area that has been identified as being involved in the process of externalization, as evidenced by fMRI. During the stimulation, participants will be engaged in a computer-based externalization task.
Procedure: High-definition transcranial direct current (HD-tDCS), placebo condition — Participants will receive a session of placebo HD-tDCS, which will be delivered following the same procedures as active HD-tDCS but the intensity of the current will be set at 2mA during the 30 first seconds at the beginning of the 25-min period of the stimulation, and equal to 0 mA for the reminding period of stimulation to simulate the tingling sensation often experienced by individuals during active stimulation.
  The placement of electrodes will be determined to specifically target the brain area that has been identified as being involved in the process of externalization, as evidenced by fMRI. During the stimulation, participants will be engaged in a computer-based externalization task

SUMMARY:
The distinction between self-generated and external information is impaired in patients with schizophrenia, who are assumed to confuse imagination with real perceptions. To better understand the underlying mechanisms of these abnormalities, the investigator will investigate the brain mechanisms supporting auditory externalization. Auditory externalization is the ability to perceive whether a sound comes from inside or outside oneself. Our study, in healthy participants, will use functional brain imaging to identify the brain areas involved in the externalization of sound sources and to test whether neuromodulation of this area can modify this ability and provide a therapeutic lead in pathological populations

DETAILED DESCRIPTION:
30 healthy participants will be included. The participants will undergo three separate visits. During the first one, the participants will listen to sounds coming from either internal or external sources while undergoing an fMRI session. This will allow us to identify the brain region involved in externalizing abilities with the highest activity. In the second and third visits, this specific region will be targeted by HD-tDCS (a non-invasive high-definition neuromodulation technique whose precision is enhanced by individual data) to modulate its activity and test its causal involvement in externalization processes. Each participant will receive both active and placebo stimulation, with the order counterbalanced. During the stimulation, participants will complete an externalization task, followed by a reality monitoring task and a self-agency task. Additionally, the investigator will gather socio-demographic and psychometric data.

ELIGIBILITY:
Inclusion Criteria:

* Having given their written informed consent
* Affiliated with a social security scheme
* French speakers and readers

Exclusion Criteria:

* With contraindication to HD-tDCS stimulation or fMRI
* With a history of or current hearing problems, including tinnitus
* Taking medication (except contraceptives)
* With a history of or current psychiatric diagnosis (DSM-5 criteria)
* First-degree relatives with a diagnosis of schizophrenia spectrum disorder or bipolar disorder (DSM5)
* Have a personal history of neurological disorders or head trauma with loss of consciousness
* With an intellectual disability (Raven's Matrices)
* With developed musical abilities (i.e., regular practice of a musical instrument for at least 10 years with assiduity or at a music school or conservatory)
* Pregnant or nursing
* Being in a period of exclusion and/or having exceeded the annual indemnity ceiling (€4,500) for other clinical research.
* Under guardianship

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-01-16 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Externalization abilities | one year
  proportion of sounds perceived as coming from an external source in the externalization task (range 0-100%)

SECONDARY OUTCOMES:
Reality monitoring performance | one year
  Scores obtained at the reality monitoring task (Brunelin et al., 2006) (accuracy, range = 0-100%)
Self-agency | one year
  Percentage of voice deviation in the self-agency task (Subramaniam et al., 2018) (pitch perturbation and variability in peak deviation in cents, cents(t) = 1200 log2 (Hertz(t )/HertzRef), mean pitch perturbation response tracks = ±100 and ± 400)
Psychometric characteristics that may influence externalization abilities and stimulation effects | baseline
  Launay-Slade Hallucinations Scale scores between 0 and 64 (LSHS; Launay and Slade)
Psychometric characteristics that may influence externalization abilities and stimulation effects | baseline
  Plymouth Sensory Imagery Questionnaire (PSIQ).Scores between 0 and 70.
Side effects of stimulation | 1 time before (baseline) and within 1 hour after stimulation
  Scores at the questionnaire on side effects of stimulation. Scores between 10 and 44 (higher scores mean worse outcome)
Mood | 1 time before (baseline) and within 1 hour after stimulation
  Mood self-questionnaire. Scores between 0 and 100 (higher scores mean worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Marine MONDINO, Phd, Principal Investigator — hospital le Vinatier
Locations (1):
- Centre Hospitalier le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided